CLINICAL TRIAL: NCT00184678
Title: Effect of Two Years of Treatment With Norditropin® SimpleXx® on Bone Mineral Density in Young Adults With Childhood-Onset Growth Hormone Deficiency
Brief Title: Effect of Growth Hormone on Bone Mineral Density in Young Adults With Child-hood Onset Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1369
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. Growth Hormone in young adults with growth hormone deficiency in childhood. This trial compares a treated group of patients with an untreated group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Child-hood onset growth hormone deficiency
* Subjects received growth hormone replacement therapy during pre-puberty and puberty

Exclusion Criteria:

* GH treatment during the month preceding randomisation
* Treatment within the previous 6 months with medication that may affect bone mineral density
* Diseases which may affect bone metabolism

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2002-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineralisation | After 2 years treatment

SECONDARY OUTCOMES:
Other markers of bone mineral content.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (29):
- Australia (4):
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Auckland
  - Novo Nordisk Investigational Site, Hamilton
  - Novo Nordisk Investigational Site, Subiaco
- Novo Nordisk Investigational Site, Graz, Austria
- Novo Nordisk Investigational Site, Brussels, Belgium
- France (3):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Marseille Cédex 05
  - Novo Nordisk Investigational Site, Toulouse
- Germany (6):
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Krefeld
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Magdeburg
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Szeged
- Novo Nordisk Investigational Site, Oslo, Norway
- Poland (5):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, Barcelona, Spain
- Novo Nordisk Investigational Site, Gothenburg, Sweden
- Switzerland (2):
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Lausanne
- United Kingdom (2):
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, London

REFERENCES:
- [Result] Zacharin M, Szarras-Czapnik M, Racz K, Keller A, Tauber M, Conway G. Growth hormone (GH) treatment improves bone mineral density during transition of GH-deficient patients from adolescence to adulthood. European Society for Paediatric Endocrinology (ESPE) 2007; Country: Finland City: Helsinki
- [Result] Zacharin M, Keller A, Chanson P, Conway G on behalf of the 1369 GHD to GHDA. Efficacy of two years' growth hormone (GH) treatment on bone mineral density in young adults with childhood-onset GH deficiency. The Endocrine Society Annual Meeting (ENDO) 2007; Country: Canada City: Toronto
- [Result] Conway G, Scarras-Czapnik M, Racz K, Keller A, Chanson P, Kappelgaard A M, Zacharin M, Hyldstrup L. Direct X-ray radiogrammetry versus dual-energy X-ray absorptiometry: assessment of bone density in young adult with childhood-onset growth hormone deficiency treated with growth hormone. The Endocrine Society Annual Meeting (ENDO) 2008; Country: USA City: San Francisco
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com